CLINICAL TRIAL: NCT06762587
Title: A Randomized, Open-Label Clinical Study on the Efficacy of Baloxavir Marboxil and Oseltamivir for Post-Exposure Prevention of Influenza in a Hospital Setting
Brief Title: Oseltamivir and Baloxavir Marboxil for Prophylaxis Against Influenza Under a Hospital-based Setting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-KY-401
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Influenza; Influenza Prophylaxis; Nosocomial Infection
Keywords: influenza; influenza prophylaxis; baloxavir marboxil; oseltamivir; nosocomial infection
MeSH Terms: conditions — Influenza, Human; Cross Infection | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baloxavir Marboxil (Experimental): Baloxavir marboxil will be administered on the first day following the close contact's enrollment in this study. Participants weighing ≤80 kg will receive 40 mg of baloxavir marboxil, while those weighing ≥80 kg will receive 80 mg.
  Interventions: Drug: Baloxavir Marboxil
- Oseltamivir Arm (Experimental): Oseltamivir will be administered once daily for 5 consecutive days following the close contact's enrollment in this study. Participants will receive 75 mg of oseltamivir once each day
  Interventions: Drug: Oseltamivir
- Control Arm (No Intervention): No antivirals will be administered to the contacts.

INTERVENTIONS:
Drug: Baloxavir Marboxil — Baloxavir marboxil will be administered on the first day following the close contact's enrollment in this study. Participants weighing ≤80 kg will receive 40 mg of baloxavir marboxil, while those weighing ≥80 kg will receive 80 mg.
  Arms: Baloxavir Marboxil
Drug: Oseltamivir — Oseltamivir will be administered once daily for 5 consecutive days following the close contact's enrollment in this study. Participants will receive 75 mg of oseltamivir once each day.
  Arms: Oseltamivir Arm

SUMMARY:
This study aims to randomly assign close contacts of hospitalized influenza virus patients to receive baloxavir marboxil prophylaxis, oseltamivir prophylaxis or no antiviral prophylaxis and monitor the incidence of clinical influenza, evaluating the prophylaxis efficiency of antivirals in a hospital setting.

DETAILED DESCRIPTION:
This study will enroll hospitalized patients diagnosed with influenza virus infection (index patients) and their roommates who are not infected with the influenza virus (close contacts). The close contacts will be randomly assigned in a 1:1:1 ratio to receive baloxavir marboxil prophylaxis, oseltamivir prophylaxis or no antiviral prophylaxis. The incidence of clinical influenza (confirmed by reverse-transcriptase polymerase chain reaction (RT-PCR) testing, along with fever and one respiratory symptom) will be monitored to evaluate the efficiency of antiviral prophylaxis in a hospital setting. The index patients will receive standard treatment for influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Index patient:
* 1. Patients or accompanying caregivers hospitalized at participating medical institutions.
* 2.The subject and/or their legal guardian both agree to participate in this clinical study, sign the informed consent form, and are able to comply with the study requirements for follow-up and completion of all study procedures and assessments.
* 3.Age ≥ 2 years.
* 4.Influenza nucleic acid positivity confirmed by throat swab, sputum and other respiratory sample through rapid antigen testing (RAT) or PCR.
* Close contact:
* 1.Patients or accompanying caregivers hospitalized at participating medical institutions.
* 2.The subject and/or their legal guardian both agree to participate in this clinical study, sign the informed consent form, and are able to comply with the study requirements for follow-up and complete all study procedures and assessments
* 3.Age ≥ 12 years.
* 4.Expected to remain hospitalized for ≥ 72 hours.
* 5.The room must contain at least one hospitalized index patient diagnosed with influenza virus within the past 72 hours, and the contact is expected to stay with the hospitalized index patient in the ward for more than 24 hours.
* 6.Throat swab on the first day tested negative for influenza virus by PCR.

Exclusion Criteria:

* Close contacts
* 1.With known allergies to the active ingredients or excipients of the investigational drug.
* 2.Close contacts diagnosed with or having experienced an influenza virus infection within the past 12 weeks.
* 3.Close contacts who have used antiviral drugs (including neuraminidase inhibitors, hemagglutinin inhibitors, and M2 ion channel blockers, such as oseltamivir, zanamivir, peramivir, favipiravir, abidol, baloxavir marboxil, amantadine, rimantadine, or any other antiviral drugs approved by NMPA) within the 2 weeks prior to screening.
* 4.Close contacts known to be pregnant or breastfeeding.
* 5. Having experienced fever (axillary temperature ≥37.3°C) in the past 3 days prior to screening.
* 6.Subjects deemed unsuitable to participate in the study by the investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Clinical Influenza within a 5-day period | up to 5 days
  Incidence of Clinical Influenza within a 5-day period is defined as the percentage of contacts who become positive for influenza based on reverse-transcriptase polymerase chain reaction (RT-PCR) testing or rapid antigen testing (RAT), along with fever (defined as axillary temperature ≥37.3℃) and at least one respiratory symptom.

SECONDARY OUTCOMES:
Incidence of influenza within a 5-day period | up to 5 days
  Incidence of Influenza within a 5-day period is defined as the percentage of contacts who become positive for influenza based on reverse-transcriptase polymerase chain reaction (RT-PCR) testing or rapid antigen testing (RAT).
Incidence of Clinical Influenza within a 10-day period | up to 10 days
  Incidence of Clinical Influenza within a 10-day period is defined as the percentage of contacts who become positive for influenza based on reverse-transcriptase polymerase chain reaction (RT-PCR) testing or rapid antigen testing (RAT), along with fever (defined as axillary temperature ≥37.3℃) and at least one respiratory symptom.
Susceptibility to antivirals by phenotyping post-baseline samples with novel mutation | up to 10 days
  Susceptibility to antivirals by phenotyping post-baseline samples with novel mutation is defined as the percentage of contacts infected with resistance-associated treatment-emergent influenza variants.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Ph.D, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No